CLINICAL TRIAL: NCT02770898
Title: Improving Family Holistic Health in Probationers- a Mixed Methods Evaluation
Brief Title: Improving Family Holistic Health in Probationers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 15-249
Record Dates: First submitted 2015-11-23; First posted 2016-05-12 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Self-efficacy; Self-esteem; Family Relationship
Keywords: probation; evidence-based; well-being; physical exercise; family well-being
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief Intervention (Experimental): The brief intervention is individual focus and consists of three main components, which include enhancing the individual personal attributes such as participant's knowledge, values, and behaviors related to physical exercise. Second, the intervention will promote changes in behavioral attributes by providing opportunities and experience in goal setting, skills development in physical exercise and self-monitoring. Finally, the brief intervention promotes family relations and well-being by encouraging individuals to share their knowledge and increase physical activities with other family members. The brief intervention will be delivered by the probation officer during regular monthly consultation.
  Interventions: Behavioral: Family Holistic Health
- Combined Intervention (Experimental): Participants allocated to the combined intervention will receive the individual brief intervention and participate in a community group program. The components in the brief intervention will also be reinforced in the group program. The group nature is designed to create an environment that is supportive of physical exercise, through role models, peer support, and encourages families to exercise with probationers.
  Interventions: Behavioral: Family Holistic Health
- Care-as-usual (No Intervention): Participants allocated to Care-as-usual arm will receive their usual services. Participants will be offered the combined interventions upon completion of 3-months follow up assessment.

INTERVENTIONS:
Behavioral: Family Holistic Health — Interventions for probationers will aim to promote physical and psychosocial health, family relationships and Family 3H (happiness, harmony and health).
  Arms: Brief Intervention; Combined Intervention

SUMMARY:
Evaluating the impact of probation on probationers is necessary for both effective practice of probation officers and their assessment of the success of their work. At present, there are limited studies that have evaluated the impact of probation services on probationers and their family. There are even fewer studies that have examined interventions on probationers' well-being and family relations in a Chinese society. Compared with the general population, probationers are associated with poorer mental (e.g., depression, lower levels of self-esteem, high level of stress) and physical health, and often experience higher levels of family conflict, and poorer quality of family relationships. Given the vulnerabilities, there is a need to strengthen and promote healthy lifestyle and enhance individual and family well-being among probationers. As part of the FAMILY project, the current study focuses on "FAMILY Holistic Health" which emphasizes a comprehensive approach to improving physical, mental, and social health and well-being. This project will be conducted as a pilot project in the Social Welfare Department (SWD) in the Eastern District of Hong Kong. Interventions will be delivered to promote and enhance probationer's wellbeing, as well as enhancing FAMILY 3Hs (Happiness, Health, and Harmony). Training programs will be provided to probation officers and/or workers of SWD in order to equip them with knowledge and skills in implementing health-related family intervention programs.

DETAILED DESCRIPTION:
To enhance individual and family well-being among probationers, family life and health education, including the skills and knowledge for physical exercise, healthy family functioning, strong communication skills, healthy interpersonal relationships, and positive self-esteem, should be strengthened and promoted. Based on the strong foundation of the FAMILY projects conducted by our research team in the past years, this project seeks to promote "FAMILY holistic health" for targeted families (i.e. probationers). The holistic health interventions are interactive and designed for behavioral changes to enhance individual well-being and encourage positive and sustainable health actions among family members. Thus, it is expected ultimately that the participants and their family members could enhance their family happiness, health, and harmony (3Hs). In sum, the project has the following contributions:

1. Strengthen evidence-based practice Hong Kong probation-related topics are scarcely studied. There is a need for rigorous studies to build and strengthen evidence-base for probation services. This study will be one of the first studies to evaluate the effectiveness of probation services on individual well-being and family well-being utilizing a mixed-methods approach.
2. Stakeholder engagement Stakeholders will be engaged throughout the research process. This promotes co-learning and empowering process, builds on strengths and resources within the community, and integrates knowledge and intervention for the mutual benefit of all partners.
3. Train-the-trainer program Training will be provided to probation officers and/or workers at the Social Welfare Department. The result of this train-the-trainers program is that front-line service workers will increase and enhance their knowledge and skills to independently and effectively carry out interventions. Probation officers will act as role models for probationers and continue to implement our knowledge and techniques in their future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Be an existing probationer with 6 months of term remaining
* Reading and writing abilities for questionnaire completion
* Have family members that are based in Hong Kong (the rationale is that one of the secondary outcome is to improve family relations)
* Probationer does not have a developmental or intellectual disability
* Probationer aged 13 and above (the rationale is that youth under 12 years of age may not have the cognitive ability to complete questionnaires)

Exclusion Criteria:

* Sexual offenders
* Drug offenders

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in Individual well-being (self-esteem, self-efficacy) | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Individual well-being will be assessed by the Rosenberg Self-esteem Scale.

SECONDARY OUTCOMES:
Physical health | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Physical health will be assessed by the SF-12v2 health survey.
Psychosocial health | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Psychosocial health will be assessed by the SF-12v2 health survey.
Behaviours on physical exercise (Adapted version of IPAC) | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Theme-related behaviours will be assessed by behavioural indicators.
Family health, happiness and harmony (3Hs) | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Family 3Hs will be assessed by the family well-being scale.
Family relations | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Family relations will be assessed by the family APGAR scale.
Satisfaction towards the program (Self-generated satisfaction scale) | T1 (baseline), T2 (one month follow-up), T3 (three months follow-up)
  Satisfaction towards the program will be assessed by a program evaluation measure.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai AY, Sit SM, Thomas C, Cheung GO, Wan A, Chan SS, Lam TH. A Randomized Controlled Trial of a Positive Family Holistic Health Intervention for Probationers in Hong Kong: A Mixed-Method Study. Front Psychol. 2021 Dec 7;12:739418. doi: 10.3389/fpsyg.2021.739418. eCollection 2021. PMID 34950083